CLINICAL TRIAL: NCT05961007
Title: A Dose Escalation Study to Evaluate the Safety and Tolerability of IBI302 Intravitreal Injection in Subjects With Neovascular Age-related Macular Degeneration and Diabetic Macular Edema AND A Multi-center, Randomized, Double-blind, Active-controlled Study to Evaluate the Efficacy and Safety of IBI302 in Subjects With Diabetic Macular Edema
Brief Title: Evaluation of IBI302 Injection in nAMD or DME
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company strategy adjustment
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI302B201
Record Dates: First submitted 2021-11-15; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Neovascular Age-related Macular Degeneration; Diabetic Macular Edema

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Masking participant and investorgastor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aflibercept (Active Comparator): only phase II
  Interventions: Drug: Intravitreal injection of Aflibercept
- IBI302 (Experimental)
  Interventions: Biological: Intravitreal injection of IBI302(dose 1); Biological: Intravitreal injection of IBI302(dose 2); Biological: Intravitreal injection of IBI302(dose 3)

INTERVENTIONS:
Biological: Intravitreal injection of IBI302(dose 1) — IBI302(dose 1) intravitreal injection given as protocol
  Arms: IBI302
Biological: Intravitreal injection of IBI302(dose 2) — IBI302(dose 2) intravitreal injection given as protocol
  Arms: IBI302
Biological: Intravitreal injection of IBI302(dose 3) — IBI302(dose 3) intravitreal injection given as protocol
  Arms: IBI302
Drug: Intravitreal injection of Aflibercept — Aflibercept intravitreal injection given as protocol
  Arms: Aflibercept

SUMMARY:
The purpose of this study is to determine the efficacy and safety of intravitreal IBI302 in the treatment of subjects with neovascular age-related macular degeneration (only in Phase I) or diabetic macular edema.

ELIGIBILITY:
Inclusion criteria

1. Willing and able to sign informed consent form and comply with visit and study procedures per protocol;
2. Male or female patiensubjects ≥ 18 yrs. of age;
3. For AMD subjects, active subfoveal or parafoveal CNV secondary to neovascular AMD; the vision decreased by nAMD;
4. For DME subjects, Type 1 or type 2 diabetes mellitus, decrease in vision determined to be primarily the result of DME in the study eye; the CST measurement of ≥ 280 μm in the study eye;
5. BCVA ETDRS letter score of 24-73 in the study eye;

Exclusion criteria

1. Concomitant diseases that may cause subjects fail to respond to the treatment or confuse the interpretation of the study results;
2. Presence of uncontrolled glaucoma in the study eye ;
3. Presence of active intraocular or periocular inflammation or infection;
4. Prior any treatment of following in the study eye:

   1. Anti-VEGF therapy or anti-complement therapy;
   2. Laser photocoagulation;
   3. History of vitreoretinal surgery;
   4. Glucocorticoid treatment(intravitreal or peribulbar) ;
5. BCVA score <19 letters in the fellow eye;
6. Anti-VEGF therapy in the fellow eye within 30 days of day 0;
7. Presence of any systemic disease: including but not limited to active infections (such as active viral hepatitis); unstable angina; cerebrovascular accident or transient cerebral ischemia (within 6 months prior to screening); myocardial infarction (within 6 months prior to screening; serious arrhythmia requiring medical treatment; liver, kidney or metabolic diseases; uncontrolled clinical disease(such as diabetes mellitus, hypertension) or malignant tumor;
8. History of severe hypersensitivity/allergy to active ingredients or any excipients of the study drug, or fluorescein and povidone iodine;
9. Pregnant or lactating women or women preparing to become pregnant or breastfeeding during the study period;
10. Participated in any clinical study of any other drug within 90 days of day 0, or attempted to participate in other drug trials during the study;
11. Other conditions unsuitable for enrollment judged by investigatiors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of ocular and non-ocular adverse events. | Up to week 20
  To evaluate the number of subjects with ocular and non-ocular adverse events, treatment emergent adverse event, adverse event of special interest, serious adverse events; number of subjects with clinical significant abnormal laboratory values, electrocardiograms (pre and post infusions), abnormal vital signs, ophthalmic and physical examinations.
DLT in each group | 7 days

SECONDARY OUTCOMES:
Change of BCVA from baseline by visit | through study completion，an average of 20 weeks
  Best corrected visual acuity (BCVA) was measured on early treatment diabetic retinopathy study(ETDRS) chart at a starting distance of 4 meters. The BCVAletter score ranges from 0 to 100(best score), and a gain in BCVA from baseline indicates an improvement in visual acuity.
Change of CST from baseline by visit | through study completion，an average of 20 weeks
  Central subfield thickness（CST） was defined as the distance between the internal limiting member and the Bruch's member using OCT, as assessed by the central reading.
Area under the concentration time curve (AUC) and Maximum plasma concentration (Cmax) | through study completion，an average of 20 weeks
The ADA and neutralizing antibody | through study completion，an average of 20 weeks
  Blood samples were obtained for measurement of anti-drug antibodies (ADAs) to IBI302 by a validated enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No